CLINICAL TRIAL: NCT06001632
Title: Changes in Muscle Strength, Inflammatory Markers, and Body Composition in Response to Alternate Day Fasting Combined With Krill Oil Supplementation in Adults With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer Human Nutrition School of Medicine, Dentistry and Nursing College of Medical, Veterinary & Life Sciences University of Glasgow, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U Glasgow
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Obesity Associated Disorder
Keywords: Obesity; Cardiometabolic risk factors; Fat mass; Fat free mass; Body composition; Muscle strength; LCn-3PUFA
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Krill oil capsules (LC n-3 PUFAs) (Experimental): 4 g/day krill oil (SuperbaBoostTM), with each 1g capsule containing 191mg EPA, 94mg DHA and 78mg choline.
  Interventions: Dietary Supplement: krill oil (SuperbaBoostTM)
- Vegetable oil capsules (Placebo Comparator): 4g/day of mixed vegetable oil (a mixture of olive oil (extra virgin, cold-pressed), maize oil (refined), palm kernel oil (refined) and medium-chain triglycerides, in the ratio 4:4:3:2).
  Interventions: Dietary Supplement: 4g/day of mixed vegetable oil

INTERVENTIONS:
Dietary Supplement: krill oil (SuperbaBoostTM) — 4 g/day of Krill oil supplements (LC n-3 PUFAs) (1g capsule containing 191mg EPA, 94mg DHA and 78mg choline).
  Arms: Krill oil capsules (LC n-3 PUFAs)
Dietary Supplement: 4g/day of mixed vegetable oil — vegetable oil capsules (mixture of olive oil (extra virgin, cold-pressed), maize oil (refined), palm kernel oil (refined) and medium-chain triglycerides, in the ratio 4:4:3:2).
  Arms: Vegetable oil capsules

SUMMARY:
The goal of this double-blind, randomised, controlled trial is to determine the effects of LC n-3 PUFAs supplementation on changes in body composition and muscle strength during body weight loss and body weight maintenance among healthy adults living with overweight and obesity. The main research questions:

* Is supplementation with LC n-3 PUFAs during dietary weight loss intervention (alternative-day fasting) attenuate the reduction in fat-free mass and muscle strength?
* Is supplementation with LC n-3 PUFAs during dietary weight loss intervention (alternative-day fasting) provide additional impact on appetite related hormones (Acylated ghrelin, GLP-1, and PYY) and cardiometabolic risk factors (Post prandial inflammatory markers and Triglycerides)? Participants will be randomly assigned to a PLACEBO (Mix-vegetables oil) or LC n-3 PUFAs group (krill oil) (1:1 basis). Both groups will follow a dietary weight loss intervention (Alternate-day fasting).

The study will last for 20 weeks that divided into 3 phases: four weeks of the preparation phase, eight weeks of body weight loss phase (Alternate Day Fasting), followed by eight weeks of body weight maintenance phase (regular diet).

DETAILED DESCRIPTION:
During the preparation phase, participants will be asked to take 4g/d krill oil capsules or placebo oil (mixed vegetable oil) with their healthy diet (their usual diet) for a period of 4 weeks. After the completion of the four weeks of the preparation phase, the weight loss intervention (Alternate Day Fasting) will start, and it last for eight weeks. Then, after the weight loss intervention, the weight maintenance phase will start, and it takes a period of 8 weeks until the end of the trial (20 weeks - study completion).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (male/female)
* body mass index (BMI) of 25 - 39.9 kg/m2
* Aged between 25 and 65 years
* stable body weight for at least three months

Exclusion Criteria:

* Smokers
* Food allergy
* On any dietary supplements or dietary regimes at the time of the study
* Participants with systolic/diastolic <90/60 mmHg and >140/90 mmHg

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in fat-free mass | 4 weeks, 12 weeks, and 20 weeks
  To assess the effect of supplementation with LCn-3 PUFA during caloric restriction on the changes of fat-free mass.
  The changes in fat-free mass will be measured by using a deuterium oxide water (D2O) technique. This technique has been used for the past 50 years to estimate total body water (TBW), which is then used to calculate fat-free mass (FFM) in kg.
  The investigators will take two saliva samples from participants in each visit.
Muscle function by Handgrip strength | 4 weeks, 12 weeks, and 20 weeks
  The Jamar hydraulic Hand dynamometer, which is a portable instrument used in clinical and research settings to precisely measure grip strength and hand function, will be used to measure handgrip strength. It has an adjustable handle that contains five grip position to suit different hand sizes and preferences. It measures the amount of force that a hand can squeeze around the dynamometer, which in term used to predict the overall muscle strength. The hand-held hydraulic system contains a measurement range of 0 to 200 pounds of force (0 to 90 kilograms), making it appropriate for testing hand grip strength.
  The dynamometer will be adjusted for participant's hand size. Then, the participant will be asked to perform as much grip pressure as possible for two to three seconds. The subjects will receive verbal guidance from the examiner to start and finish the grip test.
Chair rising test | 4 weeks, 12 weeks, and 20 weeks
  The chair rising test will be used to asses physical performance. The subjects will be asked to sit on a chair without armrests and perform a rising from a chair to a full standing position (standing fully erect to a straight and upright position) and then sitting down again as quickly as possible five times with recording time, with arms folded across the chest.
  The chair rising test will be based on seconds (s).
Fat mass | 4 weeks, 12 weeks, and 20 weeks
  To assess the effect of supplementation with LCn-3 PUFA during caloric restriction on the changes of fat mass.
  The changes in fat mass will be measured by using a deuterium oxide water (D2O) technique. This technique has been used for the past 50 years to estimate total body water (TBW), which is then used to calculate fat mass in kg.
  The investigators will take two saliva samples from participants in each visit.

SECONDARY OUTCOMES:
Appetite related hormone [Glucagon-like peptide 1 (GLP-1)] | 4 weeks, 12 weeks, and 20 weeks
  The effect of effect of LC n-3 PUFAs during dietary weight loss intervention on satiety hormone (GLP-1).
  The measurements of Plasma GLP-1 concentrations will be determined using the ELISA kit (Merck EMD Millipore, Millipore, Billerica, MO, USA).by All analyses will be performed according to the manufacturer's protocol and instructions.
Appetite related hormone [ Peptide YY (PYY)] | 4 weeks, 12 weeks, and 20 weeks
  The effect of effect of LC n-3 PUFAs during dietary weight loss intervention on satiety hormone (PYY).
  The measurements of Plasma PYY concentrations will be determined using ELISA kit (Merck EMD Millipore, Millipore, Billerica, MO, USA).
  All analyses will be performed according to the manufacturer's protocol and instructions.
Appetite related hormone [ Acylated Ghrelin] | 4 weeks, 12 weeks, and 20 weeks
  The effect of effect of LC n-3 PUFAs during dietary weight loss intervention on hunger hormone (Acylated Ghrelin).
  The measurements of Plasma Acylated Ghrelin concentrations will be determined using ELISA kit (Merck EMD Millipore, Millipore, Billerica, MO, USA).
  All analyses will be performed according to the manufacturer's protocol and instructions.
Cardiometabolic risk factor (Triglycerides) | 4 weeks, 12 weeks, and 20 weeks
  Plasma concentration of Triglycerides levels will be determined using an enzymatic hexokinase assay (Randox Laboratories Ltd., Crumlin, UK).
Cardiometabolic risk factor (Insulin) | 4 weeks, 12 weeks, and 20 weeks
  ELISA kits (Thermo Fischer, Vienna, Austria) will be used to measure concentrations of plasma insulin (Mercodia AB, Uppsala, Sweden).
Cardiometabolic risk factor (Glucose) | 4 weeks, 12 weeks, and 20 weeks
  Glucose levels will be determined using an enzymatic hexokinase assay (Randox Laboratories Ltd., Crumlin, UK).
  HOMA-IR values will be calculated using the equation developed by Matthews and colleagues (Matthews, 1985).

CONTACTS AND LOCATIONS:
Overall Officials: Mansour Alblaji, Principal Investigator — Human Nutrition School of Medicine, Dentistry and Nursing, University of Glasgow
Locations (1):
- University of Glasgow, New Lister Building, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study will published in scientific journal upon finished

REFERENCES:
- [Derived] Alblaji M, Gray SR, Almesbehi T, Morrison DJ, Malkova D. Benefits of Krill Oil Supplementation During Alternate-Day Fasting in Adults With Overweight and Obesity: A Randomized Trial. Obesity (Silver Spring). 2025 Sep;33(9):1694-1703. doi: 10.1002/oby.24354. Epub 2025 Jul 16. PMID 40671417